CLINICAL TRIAL: NCT00543179
Title: Treatment of the Dumping Syndrome With Lanreotide Autogel®
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007/064
Record Dates: First submitted 2007-10-11; First posted 2007-10-12 (Estimated); Last update posted 2007-10-12 (Estimated); Status verified 2007-10

CONDITIONS: Dumping Syndrome
MeSH Terms: conditions — Dumping Syndrome | interventions — lanreotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Somatuline (Lanreotide Autogel®)

SUMMARY:
Background Somatostatin and octreotide LAR (long-acting analogue) exert a number of inhibitory effects: on gut hormones, but also on gastro-intestinal secretion and motility.

Somatostatin analogues are effective in preventing symptoms and signs of both early and late dumping as demonstrated previously. However, octreotide LAR causes gastrointestinal side effects and the injection solution is difficult to prepare. Recently, a new somatostatin analogue with a prolonged release formulation, Lanreotide autogel (L-autogel), has become available. It is a viscous aqueous gel, composed solely of water and lanreotide. Deep subcutaneous administration may lead to increased treatment acceptance compared with intramuscular depot preparations. It is more easy to prepare and is though to cause less local side effects and technical problems than octreotide LAR. Recent studies have been done to measure the efficacy and safety of L-autogel in acromegalic treated previously with octreotide LAR. These studies showed that L-autogel is effective and well-tolerated in these patients, with equivalent or better disease control and less gastrointestinal adverse events. Until now, there is no data available on the effectivety of L-autogel in patients with a dumping syndrome. Therefore, this study aims to establish the effectiveness and tolerability of L-autogel in patients with a dumping syndrome, previously treated with octreotide LAR.

ELIGIBILITY:
Inclusion Criteria:

* Patients with typical early dumping symptoms after gastric surgery are selected on the basis of the clinical diagnostic index devised by Sigstad. In addition their dumping score after an oral glucose challenge (dumping provocation test) is positive (1,2);
* Patients with late dumping are selected on the basis of a history suggestive of postprandial hypoglycaemia, a plasma glucose of less than 3.0 mm/l at least 60 min after ingestion of 50 g glucose/ m² body surface and hypoglycaemic symptoms at least 60 min after the oral glucose load;
* Patients will be on long term octreotide LAR therapy;
* Over 18 years of age;
* Written informed consent

Exclusion Criteria:

* patients with disorders of the endocrine system, patients with severe kidney, liver or cardiovascular disease;
* Current or planned pregnancy or lactation;
* Gastrointestinal surgery one year prior to inclusion;
* Other gastrointestinal diseases that might influence symptoms of the dumping syndrome.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2007-10

PRIMARY OUTCOMES:
Responses to the dumping provocation test. Effectiveness is defined as a heart rate increase of ≤ 10 beats/min and a negative breath-hydrogen test after glucose provocation test. | baseline versus day 119

CONTACTS AND LOCATIONS:
Overall Officials: Jan BMJ Jansen, MD, PhD, Principal Investigator — UMC. St. Radboud Medical Center
Locations (1):
- UMC St. Radboud Medical Center, Nijmegen, Gelderland, Netherlands